CLINICAL TRIAL: NCT03330314
Title: An Open Label, Fixed-Sequence, Glucose Clamp Study to Compare Molar Potency of HM12460A and Insulin Glargine in Healthy Subjects
Brief Title: Molar Potency Study of HM12460A in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-INS-103
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Intravenous (IV) infusion
  Interventions: Biological: HM12460A
- Part 2: Cohort A (Experimental): Intravenous (IV) infusion (Dose A)
  Interventions: Biological: HM12460A
- Part 2: Cohort B (Experimental): Intravenous (IV) infusion (Dose B)
  Interventions: Biological: HM12460A
- Part 2: Cohort C (Experimental): Intravenous (IV) infusion (Dose C)
  Interventions: Biological: HM12460A

INTERVENTIONS:
Biological: HM12460A — HM12460A is a long-acting insulin

SUMMARY:
This is a phase 1 study to assess and compare molar potency of HM12460A and glargine in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant and non-lactating
* Males must be surgically sterile or using an acceptable contraceptive method

Exclusion Criteria:

* History of any major surgery within 6 months prior to screening
* Use of any new prescription or non-prescription drug in the last 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Blood glucose assessment of HM12460A and insulin glargine over the entire dosing period | 1 month
  - Comparison of HM12460A to insulin glargine based on blood glucose profile generated by intravenous infusion

SECONDARY OUTCOMES:
Cmax of HM12460A | 1 month
  - Maximum concentration of HM12460A over the entire dosing period
AUC of HM12460A | 1 month
  - Area Under the Curve of HM12460A over the entire dosing period

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Investigative Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided